CLINICAL TRIAL: NCT05153369
Title: Personalized and Pragmatic Three-level Model of DBT-informed Care for Youth With and/or at Familial Risk for Bipolar Disorder
Brief Title: Three-level Model of DBT-informed Care for Youth With and/or at Familial Risk for Bipolar Disorder (DB3)
Acronym: DB3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Benjamin Goldstein, Director of the Centre for Youth Bipolar Disorder, Clinician-Scientist, Professor of Psychiatry, Pharmacology & Toxicology, and Psychological Clinical Science, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 009/2021
Record Dates: First submitted 2021-11-05; First posted 2021-12-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder
Keywords: Youth; Dialectical Behavior Therapy (DBT); Psychotherapy
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: This study is targeted toward youth with and/or at familial risk for BD who, at intake, do not want and/or require full DBT. Participants will be enrolled into Level 1 - Enhanced Care or Level 2 - DBT Skills Training; for those whose circumstances change during the course of the study, such that they want and/or require full dose DBT, the intervention also includes potential dose escalation up through Level 3 - DBT Full Intervention. As the levels escalate, frequency of therapy sessions and contact with study therapist will increase. Dosing decisions will be driven by a combination of risk indicators and symptom severity, with an emphasis on emotional dysregulation, suicidality, and functional impairment, along with patient preference. Participants who are initially enrolled into Levels 1 or 2 will be able to escalate to Level 3 up until the end of their first year of enrollment. This is to ensure that they will have time to receive one full year of the DBT intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level 1 (Experimental): At enrollment, participants will be categorized according to the following criteria related to suicidality, emotion dysregulation, risk behaviors, and participant preference: No lifetime suicidal behaviors on the Columbia-Suicide Severity Rating Scale (C-SSRS) AND no active suicidal ideations with method/plan/intent in the past month on the C-SSRS (cannot score 'yes' on items > 3).
  Interventions: Behavioral: Enhanced Care
- Level 2 (Experimental): At enrollment, participants will be categorized according to the following criteria related to suicidality, emotion dysregulation, risk behaviors, and participant preference: No non-suicidal self-injurious (NSSI) behaviors in the past 3 months on the C-SSRS AND no suicide attempts (actual, interrupted and/or aborted) in the past year on the C-SSRS AND no preparatory act or behavior in the past year as measured by the C-SSRS OR participant preference.
  Interventions: Behavioral: DBT Skills Training
- Level 3 (Experimental): At enrollment, participants will be categorized according to the following criteria related to suicidality, emotion dysregulation, risk behaviors, and participant preference: NSSI behaviors in the past 3 months on the C-SSRS OR at least 1 suicide attempt in the past year (actual, interrupted, and/or aborted) on the C-SSRS OR at least 1 preparatory act or behavior in the past year as measured by the C-SSRS OR Meets youth threshold for at least 2 impulsive behavior categories on question #4 from the Structured Interview for DSM-IV Personality Disorders Borderline Personality Disorder (SIDP-IV) or 1 category is identified as severe OR participant preference during the course of treatment.
  Interventions: Behavioral: Dialectical Behavior Therapy Full Intervention

INTERVENTIONS:
Behavioral: Enhanced Care — Enhanced care aims to educate participants about bipolar disorder using a didactic approach, in addition to teaching and practicing DBT skills in an applied and relevant manner based on the participant's needs. Participants will receive a total of four sessions (approx. 60 minutes in duration), to occur once a month, at a minimum. The content will be split up into psychoeducation (2 sessions) and selected DBT skills (2 sessions). Psychoeducation will be specific to youth bipolar disorder, covering topics such as symptoms of depression and hypo/mania, medications used to treat bipolar disorder, the role of biology and the environment in emotions, and vulnerability and protective factors to emotion dysregulation and mood episodes. The content of skills sessions will be individualized and based on participant needs and goals (e.g., learning and applying skills to optimize their overall functioning, address problem behaviors and/or stressors, and/or maintain commitment to treatment).
  Arms: Level 1
Behavioral: DBT Skills Training — In DBT Skills Training, participants will only receive skills training and can choose to do this individually and/or with their individual family unit by including their parent(s) and/or sibling(s). Participants will receive 20-25 sessions (approx. 60 minutes in duration), to occur at least biweekly. Skills training will include the five standard youth DBT modules: psychoeducation about DBT and bipolar disorder, mindfulness, distress tolerance, emotion regulation, interpersonal effectiveness, and walking the middle path. The primary focus of the skills training is to impart knowledge and acquire and strengthen pragmatic skills to replace dysfunctional behaviors. If participants choose to include their family members, they will be encouraged to coach one another in effective use of skills.
  Arms: Level 2
Behavioral: Dialectical Behavior Therapy Full Intervention — The DBT full intervention is based on Miller et al.'s DBT for suicidal youth, with modifications for youth with BD. DBT will be conducted over 1 year with approximately 40-50 sessions. Sessions will alternate between individual and skills training sessions. Family involvement in skills training will be strongly encouraged, however will be up to the participant to decide. Participants in Level 3 will complete diary cards tailored for this population, assessing daily mood, suicidality, sleep, and medication adherence. Participants will report use of specified DBT skills on the diary card, and individualized treatment goals will be incorporated into the diary card (e.g., alcohol use). In addition, Level 3 will include skills coaching by phone (via phone and/or text). These brief, structured calls and/or texts function to promote skills generalization by helping the participant and any participating family member(s) use skills to achieve goals and solve problems.
  Arms: Level 3

SUMMARY:
This study seeks to bridge the knowledge-to-action gap regarding psychosocial treatment "dosing" for youth with and/or at familial risk for bipolar disorder (BD). In psychiatry, pragmatic collaborative decisions between patient and care provider about pharmacological titrations and tapers are common. Less frequently are there considerations made regarding the pragmatic dosing of psychosocial interventions. Whereas some youth clearly require full/"high-dose" treatment, others may benefit from "lower-dose" interventions, alongside re-evaluation of dosing needs over time. Furthermore, there is a subset of youth who do not require or do not want the intensity and frequency of treatment that current interventions provide. This research presents a unique opportunity to better understand different levels of care within a subspecialized outpatient mental health clinic serving youth with and/or at familial risk for BD who vary greatly in terms of risk indicators, type and severity of symptoms, associated distress, and compounding functional impairment.

DETAILED DESCRIPTION:
Bipolar disorder (BD) in adolescence is associated with poor outcomes, including impaired psychosocial functioning, substance use, and suicidality. Preliminary data using DBT as a treatment for youth BD shows improvement in depression symptoms and suicidality. At the same time, the reality is that BD is a chronic disease, and it stands to reason that a pragmatic, adaptive management approach is warranted. Developing a multi-level DBT-informed approach is advantageous for a number of reasons, in particular because this approach embraces clinical heterogeneity within and between individuals. Whereas some youth clearly require full/"high-dose" treatment, others may benefit from judicious use of "lower-dose" interventions, alongside re-evaluation of dosing needs over time. Furthermore, there is a subset of youth who do not require and/or do not want the intensity and frequency of treatment that current interventions provide. Thus far, the leading evidence-based psychosocial treatment studies in the field of youth BD have taken an "all or nothing" approach and have only been studied at one dosing level. While such an approach has certain advantages, it lacks person-centered consideration regarding pragmatic dosing. This study endeavors to determine the feasibility and effectiveness of a multi-level treatment model with dosing decisions driven by a combination of risk indicators and symptom severity (with an emphasis on emotional dysregulation, suicidality, and functional impairment; key treatment targets in dialectical behavior therapy), along with patient preference. This study proposes to implement three intensity levels of dialectical behavior therapy (DBT)-informed intervention that differ in regards to the number and frequency of sessions, parental involvement, and treatment components. This research will seek to understand the outcomes of three different levels of therapy and will examine what factors lead to the escalation of DBT dosing levels in this population.

ELIGIBILITY:
Inclusion Criteria:

1) English-speaking; 2) Age 13 years, 0 months to 23 years, 11 months; 3) Meet diagnostic criteria for BD by KSADS-PL (< 20 years of age) or SCID-5-RV (≥ 20 years of age) OR have a biological parent/sibling with BD (type I or II) confirmed via KSADS-PL or SCID-5-RV; 4) If BD-I, taking ≥1 mood stabilizing medication (i.e., antimanic anticonvulsant, antipsychotic, and/or lithium); 5) Followed by a psychiatrist who provides ongoing care; 6) Able and willing to give informed consent/assent to participate.

Exclusion Criteria:

1) Evidence of mental retardation, moderate to severe autism spectrum disorder, or organic central nervous system disorder by the K-SADS-PL (< 20 years of age), parent report, medical history, or school records that would interfere with active participation in DBT; 2) A life-threatening medical condition requiring immediate treatment; 3) Current victim of sexual or physical abuse; 4) Current substance use disorder other than mild cannabis or alcohol use disorder; 5) Meets assessment criteria for Level 3 at enrollment.

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | Baseline to 6 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 6 months to 12 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 12 months to 18 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 18 months to 24 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | Baseline to 3 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 3 months to 6 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 6 months to 9 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 9 months to 12 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 12 months to 15 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 15 months to 18 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 18 months to 21 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in symptoms using the Mood and Feelings Questionnaire (MFQ) | 21 months to 24 months
  Self-reported and parent reported depressive and manic symptoms will be measured via the Mood and Feelings Questionnaire (MFQ). Responses are made on a 3-point scale ("0=not true", "1=sometimes true" and "2=true").
Change in suicidality Suicidal Ideation Questionnaire (SIQ) | Baseline to 3 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 3 months to 6 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 6 months to 9 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 9 months to 12 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 12 months to 15 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 15 months to 18 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 18 months to 21 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 21 months to 24 months
  Youth participants will complete the self-report Suicidal Ideation Questionnaire (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | Baseline to 6 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 6 months to 12 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 12 months to 18 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 18 months to 24 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to 6 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months to 12 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 12 months to 18 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 months to 24 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | Baseline to 3 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 3 months to 6 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 6 months to 9 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 9 months to 12 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 12 months to 15 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 15 months to 18 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 18 months to 21 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 21 months to 24 months
  Youth participants will complete the Difficulties in Emotion Regulation Scale (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Treatment Satisfaction Questionnaire (18-item) | 3 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 6 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 9 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 12 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 15 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 18 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 21 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 24 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in affective lability using the Children's Affective Lability Scale (CALS) | Baseline to 3 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 3 months to 6 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 6 months to 9 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 9 months to 12 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 12 months to 15 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 15 months to 18 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 18 months to 21 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in affective lability using the Children's Affective Lability Scale (CALS) | 21 months to 24 months
  The Children's Affective Lability Scale (CALS) is a reliable 20-item adolescent- and parent-reported measure of mood lability, derived from the adult Affective Lability Scale that was specifically designed for adults with BD. It yields a total score as well as an angry/depressed factor and a disinhibited/impersistent factor. Total scores can vary from 0 to 80, with lower scores indicating a lesser degree of affective lability.
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | Baseline to 3 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 3 months to 6 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 6 months to 9 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 9 months to 12 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 12 months to 15 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 15 months to 18 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 18 months to 21 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 21 months to 24 months
  Youth participants will complete the DBT Ways of Coping Checklist (DBT-WCCL), a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Childhood Trust Events Survey (CTES) | Baseline
  Youth will complete the CTES long-form, adolescent version, a 30-item self-report screening survey that assesses exposure to adversity across a breadth of domains including physical, emotional, and sexual abuse; alcohol/drug users in home; family members in prison; caregiver with mental illness; domestic violence; loss/separation from caregiver; and other traumatic events. In addition, the CTES queries the age and perceived intensity of each type of adversity. Parents will complete the caregiver version of the CTES, a 26-item survey that asks if their child has been exposed to the same domains of adversity as queried in the adolescent version.
Number, frequency, and type of therapy sessions | At the end of study completion (5 years)
  The Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the study therapist after each therapy session.

SECONDARY OUTCOMES:
Adherence score for DBT booster sessions measured using a modified version of the Dialectical Behavior Therapy Adherence Checklist - Individual Therapy | At the end of study completion (five years)
  Video recordings will be rated for adherence using a modified version of the Dialectical Behavior Therapy Adherence Checklist - Individual Therapy (DBT AC-I) [54]. The 12 DBT strategy domains will be rated as yes/no: 1) structural strategies; 2) problem assessment strategies; 3) problem solving strategies; 4) contingency management strategies; 5) exposure strategies; 6) cognitive modification strategies; 7) validation strategies; 8) reciprocal communication strategies; 9) irreverent communication strategies; 10) dialectical strategies; 11) case management strategies; 12) protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No